CLINICAL TRIAL: NCT05342051
Title: The Effects of Immersion in 42℃ Radon, Natrium, Calcium, Bicarbonate Content Thermal-mineral Water on Chronic Low-back Pain. Controlled, Follow-up Study
Brief Title: The Effects of Immersion in 42℃ Thermal-mineral Water on Chronic Low-back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Polyclinic of the Hospitaller Brothers of St. John of God, Budapest (Other)
Responsible Party: Principal Investigator, Tamas Gati, Principal Investigator, Polyclinic of the Hospitaller Brothers of St. John of God, Budapest
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RudasCLP
Record Dates: First submitted 2022-04-07; First posted 2022-04-22 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Chronic Low-back Pain
Keywords: low back pain; Balneotherapy; spa therapy
MeSH Terms: conditions — Low Back Pain | interventions — Balneology

STUDY DESIGN:
Intervention Model Description: immersion in radon, calcium, natrium, bicarbonate content 42 ℃ thermal-mineral water 15 times in 3 weeks, plus usual care. The total mineral substance of the water is 1530 mg/l. The suggested daily time spent in water is 20 minutes altogether with breaks.
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- balneotherapy group (Experimental): balneotherapy plus usual care
  Interventions: Other: balneotherapy
- control group (No Intervention): usual care

INTERVENTIONS:
Other: balneotherapy — immersion in radon, calcium, natrium, bicarbonate content 42 ℃ thermal-mineral water 15 times in 3 weeks, plus usual care. The total mineral substance of the water is 1530 mg/l. The suggested daily time spent in water is 20 minutes altogether with breaks.
  Other Names: no intervention
  Arms: balneotherapy group

SUMMARY:
In this controlled, follow-up study the effects of immersion in 42℃ radon, natrium, calcium, bicarbonate content thermal-mineral water on clinical parameters and quality of life of patients with chronic low-back pain is evaluated. The participants in the intervention group are treated with balneotherapy plus usual care, while in the control group only with usual care. The planned participants number is 120. Follow up period is 3 months.

DETAILED DESCRIPTION:
In this controlled, follow-up study the effects of immersion in 42℃ radon, natrium, calcium, bicarbonate content thermal-mineral water on clinical parameters and quality of life of patients with chronic low-back pain is evaluated. The participants in the intervention group are treated with balneotherapy plus usual care, while in the control group only with usual care. The balneotherapy takes place in Rudas Spa in Budapest, 15 times in 3 weeks. The intensity of pain in rest and during activity evaluated on Visual Analogue Scale (VAS), the Oswestry Disability Index and the Euroqol-5D is taken at week 0., at week 3. and at week 12. The planned participants number is 120. Follow up period is 3 months.

ELIGIBILITY:
Inclusion Criteria:

* outpatients suffering from non-specific chronic low back pain standing for at least 12 weeks; only slightly reduced mobility (able to admit the treatments or visits on his own or without the help of another person);
* pain intensity of low back pain during activity at least 35 on Visual Analog Scale (0-100 mm VAS); likely degenerative symptoms

Exclusion Criteria:

* severe neurological deficit associated with the lower back;
* suspected vertebral compression of osteoporotic or other aetiology;
* malignancy;
* pain due to inflammatory spinal disease;
* severe spondylolisthesis (grade 2 or above);
* balneotherapy within 3 months prior the enrollement
* steroid therapy within 1 month prior the enrollement
* and general contraindications to balneotherapy: decompensated cardiopulmonary status (unstable hypertension, earlier tromboembolia, serious arteriosclerosis obliterans, serious varicositas, etc), unbalanced endocrinological and metabolic disease, fever condition, infectious disease, extensive inflammation/injury/absence of the skin, other severe interstitial, urogenital, and other diseases, malignancy, urine and stool incontinent, decompensated psychosis and neurosis, unconsciousness, pregnancy, postoperative status, alcoholic influence, and lack of compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
The pain during activity evaluated on Visual Analogue Scale (0-100mm) | 48 hours before the measuring time
  The pain during activity evaluated on Visual Analogue Scale (0-100mm)

SECONDARY OUTCOMES:
The pain at rest evaluated on Visual Analogue Scale (0-100mm) | 48 hours before the measuring time
  The pain at rest evaluated on Visual Analogue Scale (0-100mm)
Oswestry disability index | through study completion, an average of 12 weeks
  international questionnaire specific for back pain
EuroQol 5D index and VAS | through study completion, an average of 12 weeks
  international questionnaire evaluating the quality of life
patient acceptable symptom state (PASS) | through study completion, an average of 12 weeks
  number of patients satisfied with their condition due to low back pain

CONTACTS AND LOCATIONS:
Overall Officials: Tamas Gati, MD PhD, Principal Investigator — Polyclinic of the Hospitaller Brothers of St. John of God, Budapest
Locations (1):
- Saint Cosmas Health Center of Joseph Town, Budapest, Hungary

REFERENCES:
- [Result] Balogh Z, Ordogh J, Gasz A, Nemet L, Bender T. Effectiveness of balneotherapy in chronic low back pain -- a randomized single-blind controlled follow-up study. Forsch Komplementarmed Klass Naturheilkd. 2005 Aug;12(4):196-201. doi: 10.1159/000086305. Epub 2005 Aug 29. PMID 16137981
- [Result] Kulisch A, Bender T, Nemeth A, Szekeres L. Effect of thermal water and adjunctive electrotherapy on chronic low back pain: a double-blind, randomized, follow-up study. J Rehabil Med. 2009 Jan;41(1):73-9. doi: 10.2340/16501977-0291. PMID 19197573
- [Result] Tefner IK, Nemeth A, Laszlofi A, Kis T, Gyetvai G, Bender T. The effect of spa therapy in chronic low back pain: a randomized controlled, single-blind, follow-up study. Rheumatol Int. 2012 Oct;32(10):3163-9. doi: 10.1007/s00296-011-2145-y. Epub 2011 Sep 27. PMID 21947373
- [Result] Gati T, Tefner IK, Kovacs L, Hodosi K, Bender T. Correction to: The effects of the calcium-magnesium-bicarbonate content in thermal mineral water on chronic low back pain: a randomized, controlled follow-up study. Int J Biometeorol. 2018 May;62(5):907. doi: 10.1007/s00484-018-1505-7. PMID 29464338
- [Result] Bai R, Li C, Xiao Y, Sharma M, Zhang F, Zhao Y. Effectiveness of spa therapy for patients with chronic low back pain: An updated systematic review and meta-analysis. Medicine (Baltimore). 2019 Sep;98(37):e17092. doi: 10.1097/MD.0000000000017092. PMID 31517832
- [Result] Pittler MH, Karagulle MZ, Karagulle M, Ernst E. Spa therapy and balneotherapy for treating low back pain: meta-analysis of randomized trials. Rheumatology (Oxford). 2006 Jul;45(7):880-4. doi: 10.1093/rheumatology/kel018. Epub 2006 Jan 31. PMID 16449365
- [Result] Karagulle M, Karagulle MZ. Effectiveness of balneotherapy and spa therapy for the treatment of chronic low back pain: a review on latest evidence. Clin Rheumatol. 2015 Feb;34(2):207-14. doi: 10.1007/s10067-014-2845-2. Epub 2014 Dec 23. PMID 25535198
- [Result] Forestier R, Fioravanti A, Bender T, Santos I, Erol Forestier FB, Muela Garcia A, Francon A. Crenobalneotherapy for low back pain: systematic review of clinical trials. Int J Biometeorol. 2022 Jan;66(1):13-23. doi: 10.1007/s00484-021-02188-9. Epub 2021 Oct 9. PMID 34625843
- [Derived] Tefner IK, Bender T, Kleiber J, Hodosi K, Gati T. The effects of immersion in 42℃ radon, natrium, calcium, bicarbonate content thermal-mineral water on chronic low back pain. Controlled, follow-up study. Int J Biometeorol. 2023 Mar;67(3):527-537. doi: 10.1007/s00484-023-02433-3. Epub 2023 Jan 28. PMID 36708381